CLINICAL TRIAL: NCT01075464
Title: A Phase Ib, Open-Label, Dose-Escalation Study of the Safety and Pharmacology of MEGF0444A, a Human IgG1 Antibody, in Combination With Bevacizumab and Paclitaxel in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of the Safety and Pharmacology of MEGF0444A in Combination With Bevacizumab With or Without Paclitaxel in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEF4797g; GO01328 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Solid Cancers
Keywords: Solid Tumor
MeSH Terms: interventions — parsatuzumab; Bevacizumab; Paclitaxel

ARMS (2):
- A (Experimental)
  Interventions: Drug: MEGF0444A; Drug: bevacizumab
- B (Experimental)
  Interventions: Drug: MEGF0444A; Drug: bevacizumab; Drug: paclitaxel

INTERVENTIONS:
Drug: MEGF0444A — Intravenous escalating dose
Drug: bevacizumab — Intravenous repeating dose
Drug: paclitaxel — Intravenous repeating dose
  Arms: B

SUMMARY:
This is a Phase Ib, open-label, dose-escalation study of MEGF0444A in combination with bevacizumab, and in combination with bevacizumab and paclitaxel as therapy for locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, incurable, or metastatic solid malignancy that has progressed on or failed to respond to regimens or therapies known to provide clinical benefit

Specific to Arm A:

* For patients undergoing optional or mandatory exploratory MRI, at least one tumor lesion that represents a liver, fixed peritoneal, neck, extremity, or pelvic lesion measuring >/= 3 to 10 cm (for liver lesions) or >= 2 to 10 cm (for all other lesion locations) to be used for MRI

Specific to Arm B:

* Maximum of two prior chemotherapy regimens for metastatic disease

Exclusion Criteria:

* Anti-cancer therapy within 3 weeks prior to initiation of study treatment
* Patients who had to discontinue prior bevacizumab therapy due to intolerable toxicity
* Leptomeningeal disease
* Active infection or autoimmune disease
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, or cirrhosis
* Known primary central nervous system (CNS) malignancy or untreated or active CNS metastases
* Inadequately controlled hypertension; history of hypertensive crisis or encephalopathy; congestive heart failure (New York Heart Association Class II or greater); history of myocardial infarction or unstable angina within 6 months prior to initiation of study treatment
* History of hemoptysis; evidence of bleeding diathesis or significant coagulopathy
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to initiation of study treatment
* Serious, non-healing wound, active gastrointestinal ulcer, or untreated bone fracture

Specific to Arm B:

* Known significant hypersensitivity to paclitaxel or other drugs using the vehicle cremophor
* Previous intolerance to paclitaxel
* Grade >= 2 sensory neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities (DLTs) | Days 1 to 28 of Cycle 1
Incidence, nature, and severity of adverse events | Until 90 days after last dose of study treatment

SECONDARY OUTCOMES:
Pharmacokinetic parameters including total exposure, minimum and maximum serum concentration, clearance, and volume of distribution | Following administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (5):
- United States (5):
  - Scottsdale, Arizona
  - San Francisco, California
  - Santa Monica, California
  - Tampa, Florida
  - Nashville, Tennessee